CLINICAL TRIAL: NCT06226922
Title: Risk Factors for Postoperative Nausea and Vomiting in Surgical Patients Undergoing Patient-controlled Intravenous Analgesia.
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: K5182
Record Dates: First submitted 2024-01-18; First posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Nausea and Vomiting, Postoperative
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PCIA-PONV Group: Patient-controlled intravenous analgesia (PCIA) will be used after surgery. Patients will receive dedicated follow-up. Routine bedside visits will be conducted twice daily after surgery to assess postoperative nausea and vomiting (PONV). The severity of nausea will be evaluated using the Visual Analogue Scale (VAS), where 0 indicates no nausea and vomiting, and 10 represents the most unbearable nausea and vomiting. When the PONV score is >0 or vomiting occurs, it is defined as the PCIA-PONV group.
  Interventions: Other: No intervention
- None PCIA-PONV Group: Patient-controlled intravenous analgesia (PCIA) will be used after surgery. Patients will receive dedicated follow-up. Routine bedside visits will be conducted twice daily after surgery to assess postoperative nausea and vomiting (PONV). The severity of nausea will be evaluated using the Visual Analogue Scale (VAS), where 0 indicates no nausea and vomiting, and 10 represents the most unbearable nausea and vomiting. When the PONV score is 0, it is defined as the None PCIA-PONV Group.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The purpose of this study is to identify the risk factors for postoperative nausea and vomiting (PONV) in surgical patients undergoing patient-controlled intravenous analgesia (PCIA).

DETAILED DESCRIPTION:
Our study was a retrospective study, including patients who underwent surgery at Peking Union Medical College Hospital from July 1, 2023 to October 31, 2023 and underwent PCIA. Patient characteristics, past medical history, surgical information, intraoperative medication information, postoperative analgesia follow-up information were obtained through the electronic medical record system. The patients were divided into PCIA-PONV group and non-PCIA-PONV group depending on the occurrence of nausea and vomiting during PCIA, and all patients was also divided into PCIA-POV group and non-PCIA-POV according to whether vomiting occurred. Multivariate logistic regression analysis was used to identify the risk factors for PCIA-PONV and PCIA-POV.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Hospitalized patients
* Undergoing general anesthesia during surgery

Exclusion Criteria:

* Day surgery patients
* Accepting PCIA for less than 24 hours
* Medical record information is missing or unavailable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent surgery at Peking Union Medical College Hospital from July 1, 2023 to October 31, 2023 and received patient-controlled intravenous analgesia after surgery
Sampling Method: Non-Probability Sample
Enrollment: 1371 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
PCIA-PONV | During the PCIA procedure after surgery
  Patient-controlled intravenous analgesia (PCIA) was provided after surgery and a dedicated anesthesiologist conducted follow-up. Routine bedside visits were conducted twice a day during the PCIA procedure to evaluate the patient's postoperative nausea and vomiting. The degree of nausea was evaluated using the visual analogue scale (VAS), with 0 indicating no nausea or vomiting and 10 indicating the most severe form of unbearable nausea or vomiting. When the PONV score was greater than 4 or vomiting occurs, it was defined as PCIA-PONV.

SECONDARY OUTCOMES:
PCIA-POV | During the PCIA procedure after surgery
  Patient-controlled intravenous analgesia (PCIA) was provided after surgery and a dedicated anesthesiologist conducted follow-up. Routine bedside visits were conducted twice a day during the PCIA procedure to evaluate the patient's postoperative nausea and vomiting. When vomiting occurs, it was defined as PCIA-POV.

CONTACTS AND LOCATIONS:
Overall Officials: Shen Le, PhD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No